CLINICAL TRIAL: NCT07370025
Title: The Effect of Lullaby During Bath Time on Mother-Infant Bonding, Postpartum Depression, and Parental Self-Efficacy in Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025/728
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Newborn Infant; Bonding; Self Efficacy; Postpartum Depression (PPD)
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lullaby Group (Experimental)
  Interventions: Behavioral: Maternal Lullaby Singing
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Maternal Lullaby Singing — Mothers assigned to the intervention group will receive a brief structured education on infant bathing and the emotional role of maternal voice prior to hospital discharge. Following discharge, mothers will bathe their infants at home three times per week for two consecutive weeks (total of six sessions). During each bathing session, mothers will sing a lullaby using their own voice in a calm, quiet, and distraction-free environment. The lullaby may be a traditional cultural lullaby or spontaneous melodic humming. Recorded music will not be used. Each bathing session will last approximately 10-15 minutes, with water and room temperature adjusted to recommended neonatal care standards. Mothers will be encouraged to maintain eye contact, gentle touch, and emotional engagement with the infant throughout the bath. Researcher support will be provided via live video call during sessions to ensure adherence and safety.
  Arms: Lullaby Group

SUMMARY:
This randomized, single-blind controlled trial aims to evaluate the effects of maternal lullaby singing during infant bathing on mother-infant bonding, postpartum depressive symptoms, and perceived parenting self-efficacy in mothers of healthy term infants. The postpartum period represents a critical phase for maternal psychological adjustment, during which stress, depressive symptoms, and low parenting confidence may negatively affect the quality of mother-infant interaction and bonding. Low-cost, culturally meaningful, and non-pharmacological interventions that support maternal well-being and early bonding are therefore of particular importance.

The study will be conducted with mothers who have delivered healthy term infants in a public hospital. Eligible participants will be randomly assigned to either an intervention group or a control group. Mothers in the intervention group will receive a structured bathing education and will be instructed to bathe their infants three times per week for two consecutive weeks while singing a lullaby using their own voice in a calm and quiet home environment. Live-recorded music will not be used. The intervention emphasizes sensory interaction, emotional closeness, and maternal voice as key components. Each bathing session is expected to last approximately 10-15 minutes. The control group will receive routine postpartum care without a structured lullaby-based bathing intervention.

Outcome measures include mother-infant bonding, postpartum depressive symptoms, and perceived maternal parenting self-efficacy. Data will be collected at two time points: prior to hospital discharge (within the first 24 hours postpartum) and at the end of the two-week intervention period. Validated self-report instruments will be used for all outcome assessments.

The findings of this study are expected to provide evidence on the effectiveness of a simple, culturally embedded caregiving practice in supporting maternal mental health, strengthening mother-infant bonding, and enhancing parenting confidence during the early postpartum period. Results may inform postpartum care practices, parental counseling programs, and midwife-led supportive interventions.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have had an uncomplicated pregnancy and delivery
* Mothers who are healthy enough to care for their baby
* Mothers who have suitable conditions at home to bathe their baby
* Babies born at term (≥ 37 weeks of gestation) and with stable general health after birth

Exclusion Criteria:

* Mothers with a history of serious postpartum complications (such as postpartum hemorrhage)
* Mothers diagnosed with psychiatric illness
* Mothers who are unable to participate directly in the care of their baby (due to severe disability, mandatory bed rest, etc.)
* Mothers who cannot participate in the lullaby program due to hearing impairment
* Infants who experience serious respiratory, cardiac, or neurological problems at birth or thereafter, who have a skin disease or dermatological condition that limits bathing, who have a history of admission to the neonatal intensive care unit, or who have a chronic disease or congenital anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Mother-Infant Bonding | Baseline (within 24 hours postpartum, prior to hospital discharge) and at the end of the 2-week intervention period.
  Mother-infant bonding will be assessed using the Mother-to-Infant Bonding Scale, a validated self-report instrument consisting of 19 items measuring maternal emotional attachment, affection, and closeness toward the infant. Higher total scores indicate stronger mother-infant bonding. The total score that can be obtained on the scale ranges from 19 to 95.
Postpartum Depressive Symptoms | Baseline (within 24 hours postpartum, prior to hospital discharge) and at the end of the 2-week intervention period.
  Postpartum depressive symptoms will be measured using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-report questionnaire widely used to screen for depressive symptoms during the postpartum period. Total scores range from 0 to 30, with higher scores indicating greater depressive symptom severity.
Perceived Maternal Parenting Self-Efficacy | Baseline (within 24 hours postpartum, prior to hospital discharge) and at the end of the 2-week intervention period.
  Maternal parenting self-efficacy will be evaluated using the Perceived Maternal Parenting Self-Efficacy Scale, an 18-item self-report instrument assessing mothers' confidence in infant care, mother-infant interaction, and perceived ability to manage infant behaviors. Higher scores reflect greater perceived parenting self-efficacy.
  The total score that can be obtained on the scale ranges from 18 to 72. High scores indicate that the mother feels competent in caring for and interacting with her baby.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided